CLINICAL TRIAL: NCT06139445
Title: Effect of Manual Lymphatic Drainage on Pressure Pain Threshold, Pain Tolerance, Grip and Pinch Strength, and Two-point Discrimination
Brief Title: Manual Lymphatic Drainage for Pain, Muscle Strength, and Sensation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Emine Cihan, Assistant Prof., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/25-05
Record Dates: First submitted 2023-05-25; First posted 2023-11-18 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Manual Lymphatic Drainage Effects
Keywords: Manual lymphatic drainage; pain threshold; pain tolerance; two-point discrimination; muscle strength
MeSH Terms: interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental)
  Interventions: Other: Manual Lymphatic Drainage
- Plasebo Group (Placebo Comparator)
  Interventions: Other: Plasebo Group

INTERVENTIONS:
Other: Manual Lymphatic Drainage — Manual lymphatic drainage (MLD), one of the components of complex decongestive physiotherapy, is a gentle massage technique with proven positive effects on lymphatic circulation. MLD can be applied to different parts of the body (e.g., arms, legs, neck, abdomen, and trunk), with a different technique for each region (stationary circle, scoop, pump, and rotary)
  Arms: Study Group
Other: Plasebo Group — random superficial touches not involved in any manual technique
  Arms: Plasebo Group

SUMMARY:
To evaluate the acute effect of MLD on pressure pain threshold (PPT), pain tolerance, tactile sensation, and muscle strength in healthy young adults.

healthy young adults were included in the study. Before and after MLD and plasebo touchs, the same physiotherapist performed PPT and pain tolerance measurements, muscle strength measurements with a hand dynamometer (Jamar®) and pinchmeter (Baseline®), and two-point discrimination (2PD) evaluation with an esthesiometer.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18-30 years
* Volunteering to participate in the study

Exclusion Criteria:

* Having any skin disease
* Having a history of neurological and/or orthopedic disease
* Having a significant scar or burn tissue in the upper extremity
* Having any condition that would prevent communication

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
pressure pain threshold (PPT) | 5 minutes
  PPT measurements will be performed using a 1-cm2 surface algometer.The algometer will be positioned vertically and placed on the thenar, hypothenar, mid-ulnar, and biceps regions using the marked points. Measurements will be repeated three times. The average of these three measurements will be used for analysis.
pain tolerance | 5 minutes
  pain tolerance measurements will be performed using a 1-cm2 surface algometer.The algometer will be positioned vertically and placed on the thenar, hypothenar, mid-ulnar, and biceps regions using the marked points.The highest tolerable pressure will be used in the measurement and it will be recorded.
Evaluation of Hand Grip Strength | 5 minutes
  The Jamar will be used to measure hand grip strength.Three measurements will be made at one-minute intervals, and the average values will be recorded
Evaluation Finger Pinch Strength | 5 minutes
  A pinchmeter (Baseline®) will be used to measure finger pinch strength. Three measurements will be made at one-minute intervals, and the average values will be recorded
Two-point discrimination (2PD) | 10 minutes
  This evaluation will be performed using an esthesiometer with the participants in the sitting position with their eyes closed. Evaluation will be made from the biceps medial to the elbow. The contact time of the two-point stimulation will be adjusted to be approximately 1-2 seconds, and approximately 3-5 seconds will be waited between each stimulation. The shortest distance felt between two points provided the static 2PD value

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)